CLINICAL TRIAL: NCT02161796
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, 4-way Crossover Study to Evaluate the Dose-proportionality and Pharmacokinetics of FG-4592 in Healthy Young and Elderly Male and Female Subjects
Brief Title: A Study to Evaluate the Dose-proportionality and Effects of FG-4592 in Healthy Young and Elderly Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1517-CL-0525; 2013-001044-57 (EudraCT Number)
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: PK for FG-4592; Healthy Subjects
Keywords: Phase 1; FG-4592; Age/gender comparison
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1: young male subjects (Experimental): 3x single dose of FG-4592 and a placebo
  Interventions: Drug: FG-4592; Drug: Placebo
- 2: young female subjects (Experimental): 3x single dose of FG-4592 and a placebo
  Interventions: Drug: FG-4592; Drug: Placebo
- 3: elderly male subjects (Experimental): 3x single dose of FG-4592 and a placebo
  Interventions: Drug: FG-4592; Drug: Placebo
- 4: elderly female subjects (Experimental): 3x single dose of FG-4592 and a placebo
  Interventions: Drug: FG-4592; Drug: Placebo

INTERVENTIONS:
Drug: FG-4592 — Oral
  Other Names: ASP1517,; roxadustat
Drug: Placebo — Oral

SUMMARY:
This study evaluates the concentration of FG-4592 in the blood over a certain period after the intake of different doses, and assesses the effects, the safety and the tolerability of the study drug in healthy young and elderly male and female subjects.

On Day 1 of each of 4 periods subjects receive different single doses of FG-4592 or a placebo, depending on the treatment sequence to which they are randomized. For each period the subjects remain in the clinic for 6 days (Days -2 to 4). They are discharged after all assessments are completed on Day 4 of each period, and return for an End of Study visit (ESV) between 5 and 9 days after the last assessment of Period 4.

DETAILED DESCRIPTION:
In this study eligible subjects reside in the clinic for 4 periods of 6 days (Day -2 through Day 4). Screening takes place from Day -23 through Day -3. Subjects are admitted to the clinic on Day -2 of Period 1. Within each cohort (young and elderly subjects), subjects are randomized to one of 24 treatment sequences of 4 treatment options (3 different doses of FG-4592 and placebo) and 4 periods.

On Day 1 of each period, subjects receive a single oral dose of FG-4592 or placebo followed by a 72-hour evaluation period. Subjects are discharged on Day 4, if there are no medical reasons for a prolonged stay. Each period is separated by a wash-out period of at least 10 days between dosing on Day 1 of the previous period and dosing on Day 1 of the following period. The subjects return for an end-of-study visit (ESV) 5-9 days after the last assessment of Period 4 (or after early withdrawal).

Plasma and urine samples are collected for pharmacokinetic (PK) and pharmacodynamic (PD) assessments. Safety assessments are performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* YOUNG: Subject is a healthy young male or a healthy female subject aged 18 to 45 years of age inclusive
* ELDERLY: Subject is a healthy elderly male or female subject aged 65 or above
* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control
* Male subject must not donate sperm starting at screening and throughout the study period and for 90 days after the final study drug administration
* Female subject must be either of non-childbearing potential or, if of childbearing potential, must have a negative pregnancy test at screening and Day -2 and must use 2 forms of birth control
* Female subject must not be breastfeeding at screening or during the study period and for 28 days after the final study drug administration
* Female subject must not donate ova starting at screening and throughout the study period and for 28 days after the final study drug administration

Exclusion Criteria:

* Female subject who has been pregnant within 6 months before screening or breastfeeding within 3 months before screening
* Subject used grapefruit, grapefruit juice (more than 3 x 200 mL) or orange marmalade (more than 3 times) in the week prior to admission to the clinic until ESV
* The subject is a vulnerable subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
PK after a single dose of FG-4592 measured by area under the concentration-time curve from the time of dosing extrapolated to time infinity (AUCinf), | Days 1- 4 (all periods)
PK after a single dose of FG-4592 measured by maximum concentration (Cmax) | Days 1- 4 (all periods)

SECONDARY OUTCOMES:
PK of FG-4592 in plasma | Days 1 - 4 (all periods)
  area under the concentration-time curve (AUC) from time point 0 to time point 24 hours (AUC0-24h), unbound AUC from time point 0 to time point 24 hours (AUC0-24h,u), AUC from the time of dosing to the last measurable concentration (Clast) (AUClast), unbound AUC from the time of dosing to Clast (AUClast,u), unbound AUC extrapolated to infinity (AUCinf,u), maximum unbound plasma concentration (Cmax,u), apparent total body clearance after extra-vascular dosing (CL/F), unbound CL/F (CLu/F), fraction unbound (fu), time interval between the time of dosing and the first measurable concentration above LOQ in Plasma (tlag), time of the maximum concentration (tmax), terminal elimination half-life (t1/2), apparent volume of distribution during the terminal elimination phase after single extravascular dosing (Vz/F), unbound Vz/F (Vz,u/F)
PK of FG-4592 in urine | Days 1 - 4 (all periods)
  renal clearance (CLR), unbound CLR (CLR,u), CLR from time point 0 to 24 hours (CLR,0-24h), unbound CLR,0-24h (CLR,0-24h,u), cumulative amount of drug excreted unchanged into urine, from time of dosing extrapolated to time infinity (Aeinf), percent of drug excreted unchanged into urine from time of dosing extrapolated to time infinity in percent of dose (Aeinf%), cumulative amount of drug excreted unchanged into urine, from time of dosing up to the collection time of the last measurable concentration (Aelast), percent of drug excreted into urine (Aelast) from time of dosing up to the collection time of the last measurable concentration in percent of dose (Aelast%), cumulative amount of drug excreted unchanged into urine, from time of dosing up to the collection time of 24 hours (Ae0-24h), Ae0-24h in percent of dose (Ae0-24h%)
Plasma concentration of EPO, VEGF, reticulocytes and hepcidin | Days 1 - 4 (all periods)
  EPO(erythropoietin), VEGF(vascular endothelial growth factor)
Safety and tolerability of a single dose FG-4592 | Screening to ESV (5-9 days after the last assessment of Period 4 (or after early withdrawal))
  AEs, resting vital signs, safety laboratory tests, 12-lead safety ECG, mean heart rate per hour for 24-hours

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Parexel International GmbH, Berlin, Germany